CLINICAL TRIAL: NCT04436081
Title: Effects of THC-Free CBD Oil on Agitation in Patients With Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Old Dominion University (Other); Ananda Hemp, Inc. (Unknown)
Responsible Party: Principal Investigator, Hamid Okhravi, M.D., Associate Professor of Geriatrics and Director of Memory Clinic, Eastern Virginia Medical School
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RI-03368
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease; Dementia; Major Neurocognitive Disorder With Aggressive Behavior
Keywords: Agitation; Aggression; Neuropsychiatric symptoms; CBD Oil; Cannabinoids; Caregiver burden; Sleep quality; Behavioral and Psychological Symptoms of Dementia; Neurocognitive disorders; Psychomotor agitation; Cannabidiols
MeSH Terms: conditions — Alzheimer Disease; Dementia; Psychomotor Agitation; Aggression; Caregiver Burden; Sleep Initiation and Maintenance Disorders; Behavior; Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hemp-based CBD oil Gelcaps (Active Comparator): The intervention consists of 6 weeks oral administration of CBD oil Gelcaps, starting at a dosage of 15 mg twice per day with up titration to 45 mg twice per day. At any given dose, if participants develop side effects, the dosage will be reduced to the previous dose.
  Interventions: Drug: THC-free CBD Oil
- Oral placebo Gelcaps (Placebo Comparator): Participants in the control group will receive oral placebo Gelcaps that are identical in appearance to the CBD oil Gelcaps. Dosing will be identical to the intervention arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THC-free CBD Oil — Hemp-based CBD oil Gelcaps
  Arms: Hemp-based CBD oil Gelcaps
Drug: Placebo — Placebo Gelcaps
  Arms: Oral placebo Gelcaps

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, crossover trial that aims to 1) determine the efficacy of THC-free cannabidiol (CBD oil) in reducing the severity of agitation among participants and 2) determine whether THC-free CBD oil can reduce the burden on caregivers and increase the participants' quality of life.

DETAILED DESCRIPTION:
Individuals with Alzheimer's and other forms of dementia often go through a period of significant behavioral and psychological symptoms of dementia (BPSD). It is estimated that up to 90% of persons with dementia (PWD) experience behavior problems at some point. BPSDs can be challenging for both unpaid family caregivers as well as paid caregivers. Family caregivers provide the bulk of care for PWD and number over 15 million. One of the most common types of BPSDs is agitation with a prevalence of up to 87%, based on a recent systematic review. Agitation can lead to impaired daily functioning, prolongation of hospitalization, reduced time to institutionalization, and is associated with higher mortality. Additionally, agitated behavior is associated with increased injury to both patients and caregivers. Based on the 2018 Alzheimer's disease drug development pipeline report almost 70% of clinical trials related to BPSD are dedicated to agitation behavior. Finding ways to address agitation is necessary to improve overall quality of life for PWD and their caregivers. Currently, there are no medications available specifically for the treatment of BPSDs. The use of benzodiazepines, antipsychotics and mood stabilizing agents are common, but the risks and side effects often outweigh any benefits.

Several small studies have investigated the use of cannabinoids in the treatment of pathology and symptomology of Alzheimer's disease (AD), as well as treatment of the agitation component of BPSD. A handful of these studies showed that the symptoms of BPSD were decreased with the use of cannabinoids. However, due to small sample sizes, study design, and short trial duration of these studies, the efficacy of these agents on BPSD cannot be confirmed. In addition, cannabinoids have demonstrated anti-oxidant and anti-inflammatory effects, and both processes have been indicated as major contributors to the neurologic effects of AD. Some evidence exists that agitation is related to this neuroinflammatory process. This study will examine the effects of cannabinoids on the behavioral and psychological symptoms of individuals with a dementia diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Males/females over 50 years old.
* Have a diagnosis of dementia due to AD or mixed AD with another type of dementia.
* A Mini-Mental State Exam score (MMSE) between 4 and 28 inclusive.
* Presence of agitation with a Neuropsychiatric Inventory (NPI)-agitation/aggression subscore > 3.
* Participants and their informal caregivers must be fluent in English (includes reading, writing, and speech) and able to give informed consent.
* For patients treated with cognitive-enhancing medications (cholinesterase inhibitors (ChEI) and/or memantine), the dosage must be stable for at least 1 month (30 days). If the ChEI and/or memantine has been discontinued, patients may enroll after 15 days.
* Eligible caregivers must either live with the participant or have a minimum of 4 hours of daily contact with them.

Exclusion Criteria:

* Diagnosis of non-AD or non-mixed dementias.
* Very mild dementia or advanced dementia (MMSE: greater than 28 or less than 4).
* NPI-agitation-aggression score < 3.
* Having a serious or unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease which might confound assessment of safety outcomes as determined by the study physician.
* Presence or history of other serious psychiatric disorders or neurological conditions (e.g. psychotic disorders, bipolar disorder or schizophrenia).
* Current abuse of/dependence on marijuana, current drug abuse, current alcohol abuse.
* Having seizure disorders.
* Pregnant or breastfeeding
* Indication of baseline delirium as determined by the Confusion Assessment Method (CAM).
* Current use of lithium.
* Inability to swallow CBD oil softgels.
* Changes in dosage of anti-depressives within 4 weeks before randomization and during the study.
* Changes in dosage of antipsychotics or benzodiazepines within 1 week prior to randomization and during the study.
* Contraindications to CBD oil (history of hypersensitivity to any cannabinoid).
* Frequent falling due to orthostatic hypotension.
* Use of tricyclic antidepressants (TCA), fluoxetine, and/or carbamazepine. -Patients who reside in nursing homes.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in agitation and aggression. | Every two weeks for 15 weeks during study enrollment.
  Change in agitation and aggression will be measured by the Cohen-Mansfield Agitation Inventory (CMAI), a validated 29-item questionnaire to assess agitation. Each item is rated on a 7-point scale ranging from 1 "Never" to 7 "Several times per hour". Higher scores indicate greater agitation.
Change in caregiver burden. | Three times during the 15 weeks of study enrollment.
  Change in caregiver burden will be measured by the Zarit Burden Interview (ZBI), a validated 22-item questionnaire to assess caregiver burden. Each item is rated on a 5-point Likert scale that ranges from 0 "Never" to 4 "Nearly always," with the sum of scores ranging between 0-88. Higher scores indicate greater burden.
Change in the participant's quality of life. | Three times during the 15 weeks of study enrollment.
  Change in the participant's quality of life will be measured by the Quality-of-life assessment in dementia (DEMQOL-proxy), a validated 32-item questionnaire to assess the health related quality of life of people with dementia. Each item is rated on a 4-point scale ranging from 1 "A lot" to 4 "Not at all". Higher scores indicate a healthier quality of life.
Change in caregiver's quality of life. | Three times during the 15 weeks of study enrollment.
  Change in the caregiver's quality of life will be measured by the Measurement of quality of life in family carers of people with dementia (C-DEMQOL), a validated 30-item questionnaire to assess the quality of life for carers of someone with dementia. Each item is rated on a 5-point scale ranging from 1 "Completely" to 5 "Not at all." Higher scores indicate a healthier quality of life.

SECONDARY OUTCOMES:
Assessment of change in neuropsychiatric symptoms. | Three times during the 15 weeks of study enrollment.
  Assessment of change in neuropsychiatric symptoms for the participant will be measured by the Neuropsychiatric Inventory (NPI), a validated questionnaire that assesses dementia-related behavioral symptoms. The NPI examines 12 sub-domains of behavioral functioning. Each sub-domain is rated on the frequency of the symptoms using a 4-point scale with 1 "Occasionally" and 4 "Very frequently", the severity of the symptoms using a 3-point scale with 1 "Mild" and 3 "Marked", and the distress the symptom causes them on a 5-point scale with 1 "Not at all" and 5 "Very severely or extremely".
Assessment of change in cognitive skills. | Three times during the 15 weeks of study enrollment.
  Assessment of change in cognitive skills for the participant will be measured by the Mini Mental State Exam (MMSE), a validated 30-item questionnaire used to measure cognitive impairment among the elderly. A 30-item, clinician-administered assessment of orientation, attention, calculation, learning and memory, language, and visuospatial skills. Each correct response is summed to produce a total score out of 30 possible points.
The effect of CBD oil on sleep quantity measured by Fitbit | Measured on a daily basis during the 15 weeks of study enrollment.
  The effect of CBD oil on sleep quality will be measured for the participant and caregiver using the actigraphy function of fit bit. These measures include the amount of total sleep, amount of rapid eye movement (REM) sleep and the amount of deep and light sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Okhravi, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cerejeira J, Lagarto L, Mukaetova-Ladinska EB. Behavioral and psychological symptoms of dementia. Front Neurol. 2012 May 7;3:73. doi: 10.3389/fneur.2012.00073. eCollection 2012. PMID 22586419
- [Background] van der Linde RM, Dening T, Stephan BC, Prina AM, Evans E, Brayne C. Longitudinal course of behavioural and psychological symptoms of dementia: systematic review. Br J Psychiatry. 2016 Nov;209(5):366-377. doi: 10.1192/bjp.bp.114.148403. Epub 2016 Aug 4. PMID 27491532
- [Background] Kales HC, Gitlin LN, Lyketsos CG. Assessment and management of behavioral and psychological symptoms of dementia. BMJ. 2015 Mar 2;350:h369. doi: 10.1136/bmj.h369. PMID 25731881
- [Background] Okura T, Langa KM. Caregiver burden and neuropsychiatric symptoms in older adults with cognitive impairment: the Aging, Demographics, and Memory Study (ADAMS). Alzheimer Dis Assoc Disord. 2011 Apr-Jun;25(2):116-21. doi: 10.1097/WAD.0b013e318203f208. PMID 21192239
- [Background] Yaffe K, Fox P, Newcomer R, Sands L, Lindquist K, Dane K, Covinsky KE. Patient and caregiver characteristics and nursing home placement in patients with dementia. JAMA. 2002 Apr 24;287(16):2090-7. doi: 10.1001/jama.287.16.2090. PMID 11966383
- [Background] Khan SS, Ye B, Taati B, Mihailidis A. Detecting agitation and aggression in people with dementia using sensors-A systematic review. Alzheimers Dement. 2018 Jun;14(6):824-832. doi: 10.1016/j.jalz.2018.02.004. Epub 2018 Mar 20. PMID 29571749
- [Background] Cummings J, Lee G, Ritter A, Zhong K. Alzheimer's disease drug development pipeline: 2018. Alzheimers Dement (N Y). 2018 May 3;4:195-214. doi: 10.1016/j.trci.2018.03.009. eCollection 2018. PMID 29955663
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] Cohen-Mansfield J, Marx MS, Rosenthal AS. A description of agitation in a nursing home. J Gerontol. 1989 May;44(3):M77-84. doi: 10.1093/geronj/44.3.m77. PMID 2715584
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Smith SC, Lamping DL, Banerjee S, Harwood RH, Foley B, Smith P, Cook JC, Murray J, Prince M, Levin E, Mann A, Knapp M. Development of a new measure of health-related quality of life for people with dementia: DEMQOL. Psychol Med. 2007 May;37(5):737-46. doi: 10.1017/S0033291706009469. Epub 2006 Dec 19. PMID 17176501
- [Background] Smith SC, Lamping DL, Banerjee S, Harwood R, Foley B, Smith P, Cook JC, Murray J, Prince M, Levin E, Mann A, Knapp M. Measurement of health-related quality of life for people with dementia: development of a new instrument (DEMQOL) and an evaluation of current methodology. Health Technol Assess. 2005 Mar;9(10):1-93, iii-iv. doi: 10.3310/hta9100. PMID 15774233